CLINICAL TRIAL: NCT00682357
Title: Effect of Intraarticular Steroids on Bone Turnover in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11199
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Results first posted 2016-11-29 (Estimated); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis, intra articular steroids
MeSH Terms: conditions — Osteoarthritis | interventions — Methylprednisolone; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Methylprednisone 80 mg and Lidocaine 20 mg
  Interventions: Drug: Methylprednisolone and Lidocaine
- 2 (Experimental): Methylprednisolone 16 mg and Lidocaine 20 mg
  Interventions: Drug: Methylprednisolone and Lidocaine
- 3 (Placebo Comparator): Placebo and Lidocaine 20 mg
  Interventions: Drug: Placebo and Lidocaine

INTERVENTIONS:
Drug: Methylprednisolone and Lidocaine — Methylprednisolone 80 mg, intra-articular and lidocaine 20 mg
  Arms: 1
Drug: Methylprednisolone and Lidocaine — Methylprednisolone 16 mg intra-articular and lidocaine 20 mg
  Arms: 2
Drug: Placebo and Lidocaine — Placebo and lidocaine 20 mg
  Arms: 3

SUMMARY:
Oral and nasal steroids may enhance osteoporosis by suppressing bone formation. Intra-articular steroids may also suppress bone formation, however, the duration or relationship to a steroid dose has not been established. It is hypothesized that intra-articular steroids suppress bone formation transiently, returning to pretreatment levels within four weeks in subjects with osteoarthritis.

DETAILED DESCRIPTION:
Oral and nasal steroids may enhance osteoporosis by suppressing bone formation. Intra-articular steroids may also suppress bone formation, however, the duration or relationship to a steroid dose has not been established. It is hypothesized that intra-articular steroids suppress bone formation transiently, returning to pretreatment levels within four weeks in subjects with osteoarthritis. The purpose of the study is to determine if intra-articular steroids suppress markers of bone formation or resorption in osteoarthritis patients and whether these markers may be modified by Vitamin D or Dual-energy X-ray absorptiometry (DEXA) bone density status

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 years
* Male or postmenopausal female
* Diagnosis of knee osteoarthritis
* DEXA bone density done within the past 12 months
* Painful knee, visual analogue scale (VAS) > 4 of (10=worst)

Exclusion Criteria:

* Diabetes Mellitus Type I or II
* Systemic inflammatory illness
* Systemic infections which may be aggravated by steroid therapy
* No current or previous (< 3 years) biphosphate therapy
* Previous knee replacement surgery
* No current or previous Parathyroid hormone (PTH) therapy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Lindsley, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - Standard Dose: Methylprednisolone and Lidocaine: Methylprednisolone 80 mg, intra-articular and lidocaine 20 mg
- Group 2 - Low Dose: Methylprednisolone and Lidocaine: Methylprednisolone 16 mg intra-articular and lidocaine 20 mg
- Group 3 - Placebo: Placebo and Lidocaine: Placebo and lidocaine 20 mg
Period: Overall Study
Arm/Group | Group 1 - Standard Dose | Group 2 - Low Dose | Group 3 - Placebo
Started | 10 | 10 | 5
Completed | 10 | 10 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Standard Dose | Group 2 - Low Dose | Group 3 - Placebo | Total
Number analyzed (Participants) | 10 | 10 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 4 | 19
  >=65 years | 3 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 4 | 20
  Male | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Osteocalcin
Description: Change in serum markers of bone formation (osteocalcin) from Day 0 to Day 28.
Time Frame: Change from Baseline Visit to Day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 - Standard Dose | Group 2 - Low Dose | Group 3 - Placebo
Number analyzed (Participants) | 10 | 10 | 5
ng/mL | -2.18 (2.24) | -0.45 (2.90) | -1.10 (2.56)

2. Primary Outcome: Change in Serum Tartrate-resistant Acid Phosphatase 5b (TRACP-5b)
Description: Outcome represents the mean change in serum biomarkers of bone breakdown (TRACP-5b) from baseline visit to day 28.
Time Frame: Change from Baseline Visit to Day 28
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Group 1 - Standard Dose | Group 2 - Low Dose | Group 3 - Placebo
Number analyzed (Participants) | 10 | 10 | 5
U/L | -0.153 (0.457) | -0.295 (0.472) | -0.148 (0.804)

3. Secondary Outcome: Change in Testosterone
Description: Outcome represents the mean change in testosterone level from baseline visit to day 28.
Time Frame: Change from Baseline Visit to Day 28
Population: Only males randomized to Group 1 - Standard Dose were included in this analysis.
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Group 1 - Standard Dose | Group 2 - Low Dose | Group 3 - Placebo
Number analyzed (Participants) | 3 | 0 | 0
ng/dL | 0.08 (0.28) |  |

4. Secondary Outcome: Change in Serum Cortisol
Description: Cortisol levels were measured over 28 days. Outcome represents mean change in cortisol level between baseline visit and day 28.
Time Frame: Change from Baseline Visit to Day 28
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Group 1 - Standard Dose | Group 2 - Low Dose | Group 3 - Placebo
Number analyzed (Participants) | 10 | 10 | 5
mcg/dL | -1.16 (5.69) | 0.65 (4.59) | 1.30 (1.75)

ADVERSE EVENTS:
Arm/Group | Group 1 - Standard Dose | Group 2 - Low Dose | Group 3 - Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes